CLINICAL TRIAL: NCT06972407
Title: The Effect of rs7903146 Genotype on Islet GLP-1 Production in Humans
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-007701
Record Dates: First submitted 2025-05-05; First posted 2025-05-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Genetic Predisposition; Type2diabetes
Keywords: TCF7L2
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — exendin (9-39); Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects will be studied in the presence and absence of exendin 9-39 a competitive antagonist of the GLp-1 receptor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exendin 9-39 (Active Comparator): Exendin 9-39 will be infused during fasting and during a hyperglycemic clamp
  Interventions: Biological: Exendin 9-39
- Saline (Placebo Comparator): Saline will be infused during fasting and during a hyperglycemic clamp
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Exendin 9-39 — A competitive antagonist of the GLP-1 receptor
  Arms: Exendin 9-39
Other: Saline — Saline infusion will serve as an inactive comparator
  Arms: Saline

SUMMARY:
The investigators recently demonstrated that blockade of Glucagon-Like Peptide-1's (GLP-1) receptor (GLP1R) results in changes in islet function without changes in circulating GLP-1. These effects are more pronounced in people with early type 2 diabetes (T2DM) in keeping with increased expression of PC-1/3 and GLP-1 that is observed in diabetic islets. However, its regulation is at present unknown. Common genetic variation in the TCF7L2 locus (T-allele at rs7903146) arguably confers the greatest genetic risk of T2DM. It is associated with α- and β-cell dysfunction. TCF7L2 (the product of TCF7L2) was first described as the transcription factor necessary for proglucagon expression in intestinal L-cells (which secrete GLP-1). This led to speculation that TCF7L2 confers risk of diabetes via changes in circulating GLP-1. This has turned out to not be the case. This raises the possibility that these diabetogenic effects are mediated via an inability of islet GLP-1 to adapt to rising glycemia. Therefore, this experiment will determine the contribution of islet GLP-1 to the functional abnormalities of the islet associated with the TCF7L2 locus.

DETAILED DESCRIPTION:
The investigators recently demonstrated that blockade of Glucagon-Like Peptide-1's (GLP-1) receptor (GLP1R) results in changes in islet function without changes in circulating GLP-1. This supports other evidence (rodents and humans) that through the (inducible) expression of a prohormone convertase (PC-1/3), the α-cell can process proglucagon to intact GLP-1. 'Islet' or 'pancreatic' GLP-1 acts in a paracrine fashion to regulate insulin (basal and 1st phase) and glucagon secretion. These effects are more pronounced in people with early type 2 diabetes (T2DM) in keeping with increased expression of PC-1/3 and GLP-1 that is observed in diabetic islets.

Although pancreatic GLP-1 adapts to support islet function in T2DM, it is unclear if this mechanism is upregulated in prediabetes and whether it contributes to the phenotype(s) observed. There is evidence that α-cell proglucagon processing is subject to paracrine regulation by the β-cell. β-cell secretion of the signaling peptide 14-3-3-Zeta is decreased by GLP1R agonism, stimulating α-cell production of GLP-1. Common genetic variation in the TCF7L2 locus (T-allele at rs7903146) arguably confers the greatest genetic risk of T2DM4. It is associated with α- and β-cell dysfunction. TCF7L2 (the product of TCF7L2) was first described as the transcription factor necessary for proglucagon expression in intestinal L-cells (which secrete GLP-1). Does a relative absence or an inability of islet GLP-1 to adapt to rising glycemia explain the increased risk of T2DM associated with the T-allele at rs7903146? This experiment will determine the contribution of islet GLP-1 to the functional abnormalities of the islet associated with the TCF7L2 locus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the TT or CC genotype at rs7903146

Exclusion Criteria:

1. Age < 25 or > 70 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
2. CT genotype at rs7903146
3. HbA1c > 6.5%
4. Use of any glucose-lowering agents including metformin or sulfonylureas.
5. For female subjects: positive pregnancy test at the time of enrollment or study.
6. History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
7. Active systemic illness or malignancy.
8. Symptomatic macrovascular or microvascular disease.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in fasting glucose | Change in average glucose concentration between -30 min and 0 min of each study day (saline day vs. exendin 9-39 day)
  comparison of fasting glucose during saline vs. exendin 9-39 infusion
Change in fasting glucagon | Change in average glucagon concentration between -30 min and 0 min of each study day (saline day vs. exendin 9-39 day)
  comparison of fasting glucagon during saline vs. exendin 9-39 infusion

SECONDARY OUTCOMES:
Change in fasting insulin | Change in average insulin concentration between -30 min and 0 min of each study day (saline day vs. exendin 9-39 day)
  comparison of fasting insulin during saline vs. exendin 9-39 infusion
Change in first phase insulin secretion | Change in integrated insulin concentrations (area above baseline) between 0 min and 30 min of each study day (saline day vs. exendin 9-39 day)
  comparison of first phase insulin secretion during saline vs. exendin 9-39 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No